CLINICAL TRIAL: NCT04673279
Title: Long-term Persistence of Immunoglobulin G Antibodies Against Severe Acute Respiratory Syndrome Coronavirus 2 in a Vulnerable Neighbourhood in Buenos Aires, Argentina
Brief Title: Long-term COVID-19 Immune Response in a Vulnerable Neighbourhood in Argentina
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Hospital de Niños R. Gutierrez de Buenos Aires (Other); Ministerio de Salud GCBA (Unknown)
Responsible Party: Principal Investigator, ALICIA MISTCHENKO, principal investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 3545
Record Dates: First submitted 2020-12-13; First posted 2020-12-17 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Coronavirus Disease 2019
Keywords: Immunity; serology; antibody; SARS-CoV-2; COVID-19; vulnerability
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — blod samples for antibodies detection against dengue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serology — An enzyme linked immunosorbent assay (ELISA) developed and validated in Argentina which detects antibodies against two viral antigens, trimeric spike and the receptor binding domain (RBD) of the spike protein.

SUMMARY:
Between June 10t h and July 1st, a cross-sectional design study in an Argentina slum, showed a prevalence based on immunoglobuling G-class (IgG) antibodies against severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) of 53.4%. It remains unanswered whether natural infection produces sustained antibodies. The aim of this study is to evaluate the presence of IgG antibodies for Coronavirus disease 2019 (COVID-19) after 5 months in inhabitants of Barrio 31 who consented the Seroprevalence Study for COVID-19.

DETAILED DESCRIPTION:
Background Between June 10t h and July 1st, a cross-sectional design study was carried out in an Argentina slum over people, selected from a probabilistic sample of households showed a prevalence based on IgG-class antibodies against SARS-CoV-2 of 53.4%. In regarding to the persistence of these antibodies, the early data brought hope that acquired immunity was possible. But some subsequent studies have suggested that immune protection might be short-lived. The new findings show that people who survive a COVID-19 infection continue to produce protective antibodies against key parts of the virus for at least three to four months after developing their first symptoms. In contrast, some other antibody types decline more quickly.

It remains unanswered whether natural infection produces a sustained immunity that is capable of establishing herd immunity. The other health problem that Latin America faces is dengue, whose transmission, like SARS-CoV-2, is greater in areas with high population density such as vulnerable neighborhoods. In this context, the occurrence of the two diseases implies a risk, particularly in regions with several dengue serotypes where secondary and tertiary infections have been demonstrated and dengue epidemiological surveillance has been affected by the saturation of health system.

Objectives The aim of this study is to evaluate the presence of IgG antibodies for COVID-19 after 5 months in inhabitants of this slum who consented the Seroprevalence Study for COVID-19, and to evaluate those factors associated with the persistence of positive antibodies. As a secondary objective, the presence of positive IgG for dengue will be evaluated.

Methods Cross sectional study. Population of the study were inhabitants of the slum: men and women form 14 years of age or older were included. People will be invited to participated and detection of antibodies will be performed with ta serological tests, an enzyme linked immunosorbent assay (ELISA) developed and validated in Argentina which detects antibodies against two viral antigens, trimeric spike and the receptor binding domain (RBD) of the spike protein. Blood sample will be collected in a capillary tube from a finger prick taken at the doorstep of each person. Samples will be processed and analyzed at the "Hospital de Niños Doctor Ricardo Gutierrez" Virology laboratory.

Blood sample collection and epidemiological data were collected, and entered in a secure database.

Sample Size The first seroprevalence study included 426 inhabitants of 14 years or more. Considering a persistence of antibodies of 30% with a precision of 5% for a confidence interval of 95% 184 inhabitants should be included. This sample will be selected by a proportionate stratified random sampling, considering the ten sectors in which the slum is divided.

Statistical analysis Descriptive statistics of the data will be carried out according to the variables obtained. Continuous variables will be expressed as mean and standard deviation, and categorical variables as proportions. A multiple logistic regression model will be performed to evaluate the factors associated with the persistence of positive antibodies for SARS-CoV-2.

Dengue seroprevalence is determined globally and by geographic sector. R software version 4.0.2 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Men and women form 14 years of age or older who were included in the seroprevalence study and who have positive antibodies against severe acute respiratory syndrome coronavirus 2

Exclusion Criteria:

* deny consent

Ages: 14 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: inhabitants of Barrio Mugica: men and women form 14 years of age or older who were included in the first seroprevalence study carried on between Between June 10t h and July 1st, and who have positive antibodies against severe acute respiratory syndrome coronavirus 2
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
to estimate the proportion of people with positive IgG antibodies for COVID-19 who have positive IgG antibodies after 5 month of the first measurement | up to 20 weeks
  to estimate the proportion of people with positive IgG antibodies for COVID-19 who have positive IgG antibodies after 5 month of the first measurement

SECONDARY OUTCOMES:
to estimate the proportion of people with positive IgG antibodies for dengue | up to 20 weeks
  to estimate the proportion of people with positive IgG antibodies for dengue

CONTACTS AND LOCATIONS:
Overall Officials: Vanina Pagotto, MD MG, Study Chair — Hospital Italiano de Buenos Aires; Alicia Mistchenko, Phd, Principal Investigator — Hospital de Niños Ricardo Gutierrez; Silvana Figar, MD MG, Study Chair — Hospital Italiano de Buenos Aires; Andrea Gamarnick, Phd, Study Chair — National Council of Scientific and Technical Research, Argentina; Ana Maria Gomez Saldaño, MD MG, Study Chair — Salud Comunitaria Ministerio de Salud del Gobierno de la Ciudad de Buenos Aires; Lorena Luna, Study Chair — Salud Comunitaria Ministerio de Salud del Gobierno de la Ciudad de Buenos Aires; Julieta Salto, Study Chair — Salud Comunitaria Ministerio de Salud del Gobierno de la Ciudad de Buenos Aires; Magdalena Wagner Manslau, Study Chair — Salud Comunitaria Ministerio de Salud del Gobierno de la Ciudad de Buenos Aires; Fernan Quiroz, MD MG, Study Director — Ministerio de Salud del Gobierno de la Ciudad de Buenos Aires
Locations (1):
- Hospital de Niños Ricardo Gutierrez, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jordan RE, Adab P, Cheng KK. Covid-19: risk factors for severe disease and death. BMJ. 2020 Mar 26;368:m1198. doi: 10.1136/bmj.m1198. No abstract available. PMID 32217618
- [Background] Long QX, Tang XJ, Shi QL, Li Q, Deng HJ, Yuan J, Hu JL, Xu W, Zhang Y, Lv FJ, Su K, Zhang F, Gong J, Wu B, Liu XM, Li JJ, Qiu JF, Chen J, Huang AL. Clinical and immunological assessment of asymptomatic SARS-CoV-2 infections. Nat Med. 2020 Aug;26(8):1200-1204. doi: 10.1038/s41591-020-0965-6. Epub 2020 Jun 18. PMID 32555424
- [Background] Kellam P, Barclay W. The dynamics of humoral immune responses following SARS-CoV-2 infection and the potential for reinfection. J Gen Virol. 2020 Aug;101(8):791-797. doi: 10.1099/jgv.0.001439. PMID 32430094
- [Background] Wilder-Smith A, Tissera H, Ooi EE, Coloma J, Scott TW, Gubler DJ. Preventing Dengue Epidemics during the COVID-19 Pandemic. Am J Trop Med Hyg. 2020 Aug;103(2):570-571. doi: 10.4269/ajtmh.20-0480. Epub 2020 Jun 15. No abstract available. PMID 32539912
- [Background] Cardoso MR, Cousens SN, de Goes Siqueira LF, Alves FM, D'Angelo LA. Crowding: risk factor or protective factor for lower respiratory disease in young children? BMC Public Health. 2004 Jun 3;4:19. doi: 10.1186/1471-2458-4-19. PMID 15176983
- See also: 2019 Novel Coronavirus (COVID-19) Pneumonia with Hemoptysis as the Initial Symptom: CT and Clinical Features — http://dx.doi.org/10.3348/kjr.2020.0181
- See also: SARS-CoV-2 infection induces sustained humoral immune responses in convalescent patients following symptomatic COVID-19 — http://dx.doi.org/10.1101/2020.07.21.20159178
- See also: Community-level SARS-CoV-2 Seroprevalence Survey in urban slum dwellers of Buenos Aires City, Argentina: a participatory research. — https://www.medrxiv.org/content/10.1101/2020.07.14.20153858v2.full.pdf
- See also: Reductions in commuting mobility correlate with geographic differences in SARS-CoV-2 prevalence in New York City — https://doi.org/10.1038/s41467-020-18271-5
- See also: The COVID-19 pandemic should not jeopardize dengue control — https://journals.plos.org/plosntds/article?id=10.1371/journal.pntd.0008716